CLINICAL TRIAL: NCT03072186
Title: Proposal for Intraoperative Administration of Intravenous Indocyanine Green to Evaluate Position of the Optic Canal, Position of the Internal Carotid Arteries, Tumor Vascularization, and Vessel Encasement in Endoscopic Endonasal Cranial Base Surgery
Acronym: ICG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Daniel Prevedello, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016H0193
Record Dates: First submitted 2017-02-20; First posted 2017-03-07 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Skull Base Neoplasms; Skull Neoplasms; Bone Neoplasm; Neoplasms; Bone Diseases; Musculoskeletal Disease
MeSH Terms: conditions — Skull Base Neoplasms; Skull Neoplasms; Bone Neoplasms; Neoplasms; Bone Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- near-infrared light nasal endoscope used with ICG (Experimental): ICG will be administered to identify the blood supply at two distinct stages of endonasal cranial base surgery and tumor dissection: before intradural dissection and during tumor dissection.
  Interventions: Device: near-infrared light nasal endoscope used with ICG

INTERVENTIONS:
Device: near-infrared light nasal endoscope used with ICG — Using the near-infrared light nasal endoscope with ICG will identify anatomical landmarks and and tumor characteristics to provide a clear demonstration of the blood supply.

SUMMARY:
This study is being done to demonstrate the feasibility of using a nasal endoscope to perform intraoperative angiography of surgical field, with the goals to evaluate anatomical landmarks and tumor characteristics during skull base surgery and publish a technical note.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Patients undergoing an an EEA for cranial base pathology that will require any of the following will be eligible for the study: optic canal decompression, intradural tumor dissection, dissection of tumor around the internal carotid artery.

Exclusion Criteria:

* Less than 18 years of age
* History of sulfa, iodide, or penicillin allergy
* Previous anaphylactic reaction to ICG
* Women currently pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Prevedello, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Near-infrared Light Nasal Endoscope Used With ICG
Started | 23
Completed | 17
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Near-infrared Light Nasal Endoscope Used With ICG
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: ICG Fluorescence Ratio
Description: We aim to show that ICG fluorescence of the tumor intraoperatively is directly proportional to the contrast enhancement of the tumor from preoperative MRI. Enhancement is shown in ratio form on a scale of 0.01-1.00 showing enhancement ratios of 1. gland to internal carotid artery compared to blood fluorescence and 2. tumor tissue to blood fluorescence. Video recordings of intra-operative ICG fluorescence was compared to pre-operative imaging enhancements and compared in ratio format with a possible score of 0.01-1.00 The higher the ratio, the more closely the intra-operative fluorescence was related to the pre-operative imaging enhancements. 1.00 is considered to have the same enhancing brightness on pre-operative imaging as intra-operative video surveillance.
Time Frame: Before intradural dissection and during tumor dissection.
Population: Patients undergoing tumor resection via endoscopic endonasal approach. Tumor pathologies included: pituitary adenoma (10), chordoma (4), tuberculum sellae meningioma (3), chondrosarcoma (1) estesioneuroblastoma (1) and Rathke's cleft cyst (1)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Near-infrared Light Nasal Endoscope Used With ICG
Number analyzed (Participants) | 20
Ratio
  gland to internal carotid artery ratio: number analyzed (Participants) | 10
  gland to internal carotid artery ratio | 0.92 (0.001)
  tumor to internal carotid artery ratio: number analyzed (Participants) | 10
  tumor to internal carotid artery ratio | 0.82 (0.006)

ADVERSE EVENTS:
Time Frame: Patient adverse events were tracked while the patient was in the hospital. No longer than one week.
Description: Adverse events were only recorded if the event was related to the study procedure. Events that occur due to the standard of care surgery were not recorded.
Arm/Group | Near-infrared Light Nasal Endoscope Used With ICG
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT03072186/Prot_000.pdf